CLINICAL TRIAL: NCT03237039
Title: Classification of the Sagittal Profile of the Spine in Asymptomatic Elderly Subjects
Acronym: EOS60
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EOS60
Record Dates: First submitted 2017-07-19; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Aged; Asymptomatic Condition
Keywords: Roussouly type; spine alignment; fall-risk; gait cycle analysis
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Intervention Model Description: symptomatic elderly subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- X-ray examination, fall-risk and gait (Other): simultaneous acquisition in upright position of two full-body radiographic images, one in the coronal plane and one in the sagittal plane. In addition, 40 out of 160 subjects will undergo fall-risk assessment and gait cycle analysis evaluation.
  Interventions: Radiation: X-ray examination; Other: fall-risk assessment; Other: gait cycle analysis

INTERVENTIONS:
Radiation: X-ray examination — Radiological examination of frontal and lateral planes, simultaneously acquired with low dose X-ray system (EOS system, France) in one single exposition. The evaluation of the radiographic images will be performed by an orthopedic physician.Image processing will be performed by a biomedical engineer through sterEOS proprietary software and will provide the anatomical parameters needed to classify the sagittal profile.
Other: fall-risk assessment — This evaluation will be performed after the radiographic scan, in the same day. The fall-risk assessment test will be performed by a biomedical engineer through OAK device (OAK, Khymeia, Italy). The OAK device integrates two force plates and sensory elastic straps applied to pelvis and limbs. This test, which takes approximately twenty minutes, accounts eight consecutive postural equilibrium exercises and provide the automatic detection of subject's postural parameters. At the end of the test, the fall-risk rating is automatically assigned.
Other: gait cycle analysis — This assessment will be performed in the same session of fall-risk evaluation. The gait cycle analysis, which takes approximately forty minutes, will be executed by a biomedical engineer. Adhesive passive reflective markers will be placed on the skin according to a protocol suitable to characterize the alignment of lower limbs and trunk. The markers trajectories during walk will be recorded by an eight cameras optoelectronic system (BTS smart-D, Italy). A force platform (Kistler, Switzerland) placed in the middle of the pathway will detect the forces exchanged with the ground. The data analysis will provide the kinematic and kinetic descriptive parameters of gait cycle.

SUMMARY:
Principal aim The main purpose of the study is to describe the distribution of the sagittal profile in elderly subjects in order to bridge the gap present in this type of screening, evaluated in the literature for adults only (i.e. 160 subjects considered by Roussouly et al. in 2005). This classification assigns an integer value from 1 to 4 in relation to the evaluation of alignment of the lumbar spine and pelvis in the sagittal plane. The population description is therefore divided into four categories. The extension of this classification to elderly can provide useful support for the clinical evaluation and the specific treatment of the elderly patients.

Secondary aims The study aims in addition to evaluate the relation between the spine sagittal profile and the objective indexes obtained from the assessment of fall-risk and gait cycle analysis. Accordingly, a subgroup of 40 subjects out of the 160 will be evaluated. This subgroup will consider the subjects older than or equal to 74 years, where the risk of falling is most likely to be expected.

DETAILED DESCRIPTION:
Introduction:

The classification of spine sagittal profile can be an essential prediction factor for the specific prevention and treatment of patient's pathologies. Despite high variability, sagittal alignment can be accurately measured by radiographic examination and is fully replicable. To this regard, a classification of the lumbar profile and pelvis in the sagittal plane was proposed by Roussouly et al. Specifically, four different typologies can be recognized. These typologies classify the profile of the lumbar curve and are directly related to the quantification of the pelvic inclination. The study by Roussouly et al. examined 160 asymptomatic subjects aged between 18 and 45 years and confirmed the high inter-individual variability of the sagittal profile. Unfortunately, this classification has not been extended to elderly. In this regard, it has been shown that peculiar changes in the sagittal profile are particularly evident in aging, such as the advancement of the average sagittal axis and the tendency to decrease of the degree of lumbar lordosis.

According to that, extending the classification of the spine sagittal alignment in elderly results of prime importance. Furthermore, extending this classification will also provide useful information supporting the clinical evaluation and the specific treatment of elderly patients (e.g. better understanding the association between spine alignment and the development of degenerative alterations). In addition to this primary objective, this study aims to assess the relation between postural imbalance (due to alterations of the sagittal profile) and motor functionality in elderly. A subgroup of the enrolled subjects, equal to one quarter of the total size, will undergo fall-risk assessment and gait cycle analysis. This subgroup will account subjects older than or equal to 74 years, where the risk of falling is more likely to occur. The objective indices obtained from these analyses will be put in relation with the classification of the spine sagittal profile.

Aims of the study:

The primary aim of this study is to classify the spine sagittal profile in elderly asymptomatic subjects (older than or equal to 60 years) through the semi-automatic analysis of low dose radiographic images obtained through a validated radiographic system (EOS Imaging System, France). The study will evaluate 160 subjects, at least 40 of whom will have an age greater than or equal to 74 years. According to Roussouly et al., the classification of the spine alignment will assign an integer value ranging from 1 to 4, in relation to the evaluation of the lumbar spine and pelvis in the sagittal plane. Secondary aim of the study will be to investigate the relation between the classification of spine sagittal profile and the objective indexes characterizing the fall-risk and the gait cycle analysis. This assessment will take into account the subgroup of 40 subjects aged 74 years or more.

Radiographic examination:

The radiographic examination will be performed with the EOS low-dose X-ray radiation system by a radiology technician. The examination, which will take about 10 seconds, will allow the simultaneous acquisition in upright position of two full-body radiographic images, one in the coronal plane and one in the sagittal plane. The evaluation of the radiographic images will be performed by an orthopedic physician. Image processing will be performed by a biomedical engineer through sterEOS proprietary software and will provide the anatomical parameters needed to classify the sagittal profile.

Assessment of fall-risk:

This evaluation will be performed after the radiographic examination, in the same session. The fall-risk assessment test will be performed by a biomedical engineer through OAK device (OAK, Khymeia, Italy). The OAK device integrates two force plates and sensory elastic straps applied to pelvis and limbs. This test, which takes approximately twenty minutes, accounts eight consecutive postural equilibrium exercises and provide the automatic detection of subject's postural parameters. At the end of the test, the fall-risk rating is automatically assigned.

Gait cycle analysis:

This assessment will be performed in the same session of fall-risk evaluation. The gait cycle analysis, which takes approximately forty minutes, will be executed by a biomedical engineer. Adhesive passive reflective markers will be placed on the skin according to a protocol suitable to characterize the alignment of lower limbs and trunk. The markers trajectories during walk will be recorded by an eight cameras optoelectronic system (BTS smart-D, Italy). A force platform (Kistler, Switzerland) placed in the middle of the pathway will detect the forces exchanged with the ground. The data analysis will provide the kinematic and kinetic descriptive parameters of gait cycle.

Statistical analysis:

The total sample size was chosen considering the classificatory purpose of the present study and its descriptive and non-comparative intent. It was therefore considered as appropriate to match the number of 160 subjects evaluated in previous study to classify the spine sagittal alignment in adult subjects. Concerning the secondary aim of the study, the correlation between the Roussouly type (identifying the spine sagittal alignment) and the indexes characterizing fall-risk and gait cycle will be assessed. The significance of the Pearson correlation coefficient or of Spearman correlation coefficient, in case of non-Gaussian data, will be tested according to two-tailed t-test or permutation distribution test, respectively. Statistical significance will be considered at p <0.05 level. To this regard, the sample size requested to guarantee the significance (with α = 0.05 and statistical power = 95%) of a correlation value defined as 'strong' (not less than 0.6, in absolute value), is equal to 30. The number of 40 subjects planned for the secondary aim thus fulfills the requirements for the correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* older than or equal to 60 years
* subscription of informed consent

Exclusion Criteria:

* Significant painful episodes linked to the spine in the last 2 years
* Early surgical interventions involving the spine
* scoliosis or other spine pathologies (vertebral, neurological, muscular)
* Obesity (BMI> 30 kg / m2)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-04-03 (Estimated); Study Completion 2019-04-03 (Estimated)

PRIMARY OUTCOMES:
Classification of Roussouly type | Through study completion, an average of 18 months
  This classification assigns an integer value ranging from 1 to 4, in relation to the evaluation of lumbar spine and pelvis alignment in the sagittal plane. It will be acquired to describe subjects' population, and correlations with fall-risk and gait cycle indexes will be checked for.
Subject's weight | Through study completion, an average of 18 months
  Subject's weight (kg) will be acquired to describe subjects' population
Subject's height | Through study completion, an average of 18 months
  Subject's height (cm) will be acquired to describe subjects' population
Thoracic kyphosis | Through study completion, an average of 18 months
  Thoracic kyphosis (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.
Lumbar lordosis | Through study completion, an average of 18 months
  Lumbar lordosis (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.
Pelvic incidence | Through study completion, an average of 18 months
  Pelvic incidence (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.
Sacral slope | Through study completion, an average of 18 months
  Sacral slope (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.
Pelvic tilt | Through study completion, an average of 18 months
  Pelvic tilt (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.
Lateral pelvic inclination | Through study completion, an average of 18 months
  Lateral pelvic inclination (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.
Pelvic torsion | Through study completion, an average of 18 months
  Pelvic torsion (°) will be accounted for the spine alignment classification, and correlations with fall-risk and gait cycle indexes will be checked for.

SECONDARY OUTCOMES:
Fall-risk score | Through study completion, an average of 18 months
  Evaluation of the fall-risk with the OAK device (OAK, Khymeia, Italy). The device automatically evaluates the fall-risk score, an integer value ranging from 0 to 24, where 0 indicates maximum risk and 24 the minimum.
Functional forward flexion | Through study completion, an average of 18 months
  Functional forward flexion (cm) will be automatically computed by the OAK device.
CoP sway area | Through study completion, an average of 18 months
  Sway area of the center of pressure (cm2) will be automatically computed by the OAK device.
Gait analysis: stance phase | Through study completion, an average of 18 months
  Stance phase (% of total gait cycle time) will be evaluated for both the right and left legs.
Gait analysis: swing phase | Through study completion, an average of 18 months
  Swing phase (% of total gait cycle time) will be evaluated for both the right and left legs.
Gait analysis: stride length | Through study completion, an average of 18 months
  Stride length (m) will be evaluated for both the right and left legs.
Gait analysis: average walking speed | Through study completion, an average of 18 months
  Average walking speed (m/s).
Gait analysis: average step cadence | Through study completion, an average of 18 months
  Average step cadence (steps/min)
Gait analysis: maximum hip flexion | Through study completion, an average of 18 months
  Maximum hip flexion (°) will be evaluated for both the right and left hips.
Gait analysis: maximum hip extension | Through study completion, an average of 18 months
  Maximum hip extension (°) will be evaluated for both the right and left hips.
Gait analysis: maximum hip flexion moment | Through study completion, an average of 18 months
  Maximum hip flexion moment (Nm) will be evaluated for both the right and left hips.
Gait analysis: maximum hip extension moment | Through study completion, an average of 18 months
  Maximum hip extension moment (Nm) will be evaluated for both the right and left hips.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Brayda-Bruno, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- Marco Brayda-Bruno, MD, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietrich TJ, Pfirrmann CW, Schwab A, Pankalla K, Buck FM. Comparison of radiation dose, workflow, patient comfort and financial break-even of standard digital radiography and a novel biplanar low-dose X-ray system for upright full-length lower limb and whole spine radiography. Skeletal Radiol. 2013 Jul;42(7):959-67. doi: 10.1007/s00256-013-1600-0. Epub 2013 Mar 28. PMID 23536038
- [Background] Dreischarf M, Albiol L, Rohlmann A, Pries E, Bashkuev M, Zander T, Duda G, Druschel C, Strube P, Putzier M, Schmidt H. Age-related loss of lumbar spinal lordosis and mobility--a study of 323 asymptomatic volunteers. PLoS One. 2014 Dec 30;9(12):e116186. doi: 10.1371/journal.pone.0116186. eCollection 2014. PMID 25549085
- [Background] Gelb DE, Lenke LG, Bridwell KH, Blanke K, McEnery KW. An analysis of sagittal spinal alignment in 100 asymptomatic middle and older aged volunteers. Spine (Phila Pa 1976). 1995 Jun 15;20(12):1351-8. PMID 7676332
- [Background] Hammerberg EM, Wood KB. Sagittal profile of the elderly. J Spinal Disord Tech. 2003 Feb;16(1):44-50. doi: 10.1097/00024720-200302000-00008. PMID 12571484
- [Background] Jackson RP, Peterson MD, McManus AC, Hales C. Compensatory spinopelvic balance over the hip axis and better reliability in measuring lordosis to the pelvic radius on standing lateral radiographs of adult volunteers and patients. Spine (Phila Pa 1976). 1998 Aug 15;23(16):1750-67. doi: 10.1097/00007632-199808150-00008. PMID 9728376
- [Background] Jackson RP, Hales C. Congruent spinopelvic alignment on standing lateral radiographs of adult volunteers. Spine (Phila Pa 1976). 2000 Nov 1;25(21):2808-15. doi: 10.1097/00007632-200011010-00014. PMID 11064527
- [Background] Pellet N, Aunoble S, Meyrat R, Rigal J, Le Huec JC. Sagittal balance parameters influence indications for lumbar disc arthroplasty or ALIF. Eur Spine J. 2011 Sep;20 Suppl 5(Suppl 5):647-62. doi: 10.1007/s00586-011-1933-0. Epub 2011 Aug 16. PMID 21845396
- [Background] Roussouly P, Gollogly S, Berthonnaud E, Dimnet J. Classification of the normal variation in the sagittal alignment of the human lumbar spine and pelvis in the standing position. Spine (Phila Pa 1976). 2005 Feb 1;30(3):346-53. doi: 10.1097/01.brs.0000152379.54463.65. PMID 15682018
- [Background] Shah DJ, Sachs RK, Wilson DJ. Radiation-induced cancer: a modern view. Br J Radiol. 2012 Dec;85(1020):e1166-73. doi: 10.1259/bjr/25026140. PMID 23175483
- [Background] Stagnara P, De Mauroy JC, Dran G, Gonon GP, Costanzo G, Dimnet J, Pasquet A. Reciprocal angulation of vertebral bodies in a sagittal plane: approach to references for the evaluation of kyphosis and lordosis. Spine (Phila Pa 1976). 1982 Jul-Aug;7(4):335-42. doi: 10.1097/00007632-198207000-00003. PMID 7135066
- [Background] Vedantam R, Lenke LG, Keeney JA, Bridwell KH. Comparison of standing sagittal spinal alignment in asymptomatic adolescents and adults. Spine (Phila Pa 1976). 1998 Jan 15;23(2):211-5. doi: 10.1097/00007632-199801150-00012. PMID 9474728